CLINICAL TRIAL: NCT05064436
Title: A Phase 1, Open-label, Multi-part Study to Evaluate the Safety, Tolerability, Kinetics, Biodistribution, and CNS Signal of the Positron Emission Tomography Ligand 11C-BMS-986196 in Healthy Participants After Intravenous Administration and to Evaluate the Safety, Tolerability, Kinetics, and CNS Signal Repeatability of 11C-BMS-986196 After Repeat Intravenous Administration in Participants With Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability, Kinetics, Biodistribution and Repeatability of 11C-BMS-986196 After Intravenous (IV) Administration in Healthy Participants and After Repeat IV Administration in Participants With Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IM038-010; 2021-001986-19 (EudraCT Number)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis (MS); Healthy Participants; 11C-BMS-986196; PET tracer
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - Healthy Participants (Experimental)
  Interventions: Drug: 11C-BMS-986196
- Part B - Participants with MS (Experimental)
  Interventions: Drug: 11C-BMS-986196

INTERVENTIONS:
Drug: 11C-BMS-986196 — Specified dose on specified days
  Other Names: BMS-986196

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, kinetics, biodistribution and central nervous system signal of 11C-BMS-986196 after intravenous (IV) administration in healthy participants and after repeat IV administration in participants with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

For Parts A & B:

* Body mass index (BMI) of 18 to 34 kg/m2, inclusive, and total body weight ≥ 50 kg
* Documentation of normal Allen's test result at Screening and on PET scanning days in the arm that will be used for arterial line placement

For Part A only:

• Healthy male and female participants without clinically significant deviation from normal in medical history, physical examination (PE), electrocardiograms (ECGs), and clinical laboratory determinations

For Part B only:

* Male or female participant diagnosed with MS according to the 2017 revisions of the McDonald diagnostic criteria
* Expanded Disability Status Scale (EDSS) score between 0 to 6.5, inclusive, at Screening

Exclusion Criteria:

For Parts A & B:

* Benign MS defined as a baseline EDSS of 2.0 with MS diagnosis ≥ 10 years prior to Day 1. Spinal MS without clinical or radiological evidence of brain lesions. Any other combination of clinical and radiological data suggestive of an absence of inflammatory brain lesions.
* Any major surgery within 4 weeks of study treatment administration and/or any minor surgery within 2 weeks of tracer administration

For Part A only:

• Any significant acute or chronic medical illness

For Part B only:

* Any significant acute or chronic medical illness (other than MS) posing a risk to the participant's safety or negatively affecting the ability to detect CNS PET signal
* MS relapse within 14 days prior to Day 1. Participants with a MS relapse within 30 days prior to Day 1 must agree to have their second PET scan scheduled on Day 1 or Day 2

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution - 0001, Ann Arbor, Michigan, United States
- Local Institution - 0002, London, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants randomized and treated
Groups:
- Part A: BMS-986196 Approximately 370MBq, equivalent to up to 20 μg
- Part B: BMS-986196 Approximately 370 MBq, equivalent to up to 20 μg
Period: Overall Study
Arm/Group | Part A | Part B
Started | 6 | 4
Completed | 5 | 4
Not Completed | 1 | 0
Not completed — Other Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.0 (12.0) | 50.8 (4.0) | 41.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Based on Severity.
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.
Time Frame: From first visit up to 9 days post
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 4
Participants
  Mild | 1 | 1
  Moderate | 1 | 2
  Severe | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiograms.
Description: Number of participants with clinically significant changes in electrocardiograms.
Time Frame: From first visit up to 9 days post
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs.
Description: Number of participants with clinically significant changes in vital signs.
Time Frame: From first visit up to 9 days post
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Values.
Description: Number of participants with clinically significant changes in laboratory values.
Time Frame: From first visit up to 9 days post
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Phsyical Examinations.
Description: Number of participants with clinically significant changes in phsyical examinations.
Time Frame: From first visit up to 9 days post
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 4
Participants | 2 | 3

6. Primary Outcome: Number of Participants With Clinically Significant Changes in C-SSRS.
Description: Number of participants with clinically significant changes in C-SSRS.
  Columbia-Suicide Severity Rating Scale (C-SSRS).
  The entire Columbia Suicide Severity Rating Scale (C-SSRS) will be administered, but the investigators will use its' Suicidal Ideation Intensity scale (0-25 score range summed from five items, with higher scores indicating more severe suicidal ideation) as the primary outcome.
  Data Not Collected
Time Frame: Data Not Collected
Population: Study terminated before data collection for this endpoint occurred.
Arm/Group | Part A | Part B
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Radiation Dosimetry Calculated From PET-CT Images in Healthy Participants
Description: Measurement and assessment of radiation exposure and absorption of ionizing radiation in body tissue.
  The Organ Level Internal Dose Assessment (OLINDA) 2.0 software package (Hermes Medical Solutions) was used to estimate the organ and whole-body radiation absorbed doses. OLINDA uses Medical Internal Radiation Dose (MIRD) methodology (Stabin, Sparks, and Crowe 2005). The NURBs ICRP-89 adult male (73 kg) model was used to calculate the referent s-factors (Valentin and Streffer 2002). Tissue weighting factors defined in (ICRP Publication 103, 2007) were used to calculate the whole body effective dose (ED). All other MIRD assumptions about the homogeneity of source organ distribution were employed.
Time Frame: 2 hours
Population: All Treated Population
Measure: Mean (Standard Deviation); unit: uSv/MBq
Arm/Group | Part A | Part B
Number analyzed (Participants) | 5 | 0
uSv/MBq | 4.36 (0.57) |

8. Primary Outcome: Image Acquisition Window After Tracer Administration
Description: Period of time required to collect the imaging data during a scan.
  Participants received a bolus intravenous administration of up to 370 MBq of 11CBMS- 986196. Immediately following the 11C-BMS-986196 administration, dynamic PET emission data were acquired for 90 minutes in a single bed position focused on the cranium.
  For PET acquisitions, a low dose CT scan was performed before administration of the radiotracer, to enable correction for attenuation of emitted radiation.
Time Frame: 90 Mins
Population: All Treated Population
Measure: Median (Full Range); unit: Mins
Arm/Group | Part A | Part B
Number analyzed (Participants) | 5 | 4
Mins | 90 [0 to 90] | 90 [0 to 90]

9. Primary Outcome: Percentage of Participants With Test Repeatablity Based on SUV.
Description: Standardized uptake value (SUV) is Semi-quantitative measurement of tracer uptake in body tissue defined as ratio of radioactivity per unit volume of a region of interest to the radioactivity per unit volume of the whole body.
  Test-retest repeatability based on standardized uptake value (SUV) of CNS PET images in participants with MS: The test-retest repeatability will be based on a quantitative analysis of cranial PET images and will be evaluated for the Response-Evaluable 3 population. The test-retest repeatability (%), which is defined based upon the absolute value of the difference between test and retest values normalized by their mean:
  Test-Retest difference = RT-T Test-retest repeatability (%) = 100%-2×|(RT-T)/(RT+T)|×100%
  with T being the calculated value for the parameter measured at Visit 1 (test, T) and RT being the calculated value for the same parameter measured at Visit 2 (retest, RT).
Time Frame: 2 hours
Population: Response-Evaluable Population with MS, 0 participants in Part A had MS
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A | Part B
Number analyzed (Participants) | 0 | 3
percentage
  Brain-Grey Matter |  | 96.163 (3.621)
  Brain-Lesion |  | 95.930 (3.427)
  Brain-White Matter |  | 96.128 (3.670)
  Cerebellum-Grey Matter |  | 95.114 (3.557)
  Cerebellum-White Matter |  | 93.541 (6.164)
  Cerebral Cortex-Grey Matter |  | 96.601 (3.675)
  Cerebral Cortex-White Matter |  | 96.697 (3.571)
  Cerebral Subcortex-Grey Matter |  | 95.833 (2.957)
  Cerebral White Matter-White Matter |  | 95.912 (3.893)

10. Primary Outcome: Percentage of Participants With Test Repeatablity Based on VT.
Description: Volume of Distribution (VT) is the ratio of the radioligand concentration in a region of interest to the radioligand concentration in plasma at equilibrium.
  Test-retest repeatability based on VT of CNS PET images in participants with MS: The test-retest repeatability will be based on a quantitative analysis of cranial PET images and will be evaluated for the Response-Evaluable 3 population. The test-retest repeatability (%), which is defined based upon the absolute value of the difference between test and retest values normalized by their mean:
  Test-Retest difference = RT-T Test-retest repeatability (%) = 100%-2×|(RT-T)/(RT+T)|×100%
  with T being the calculated value for the parameter measured at Visit 1 (test, T) and RT being the calculated value for the same parameter measured at Visit 2 (retest, RT).
Time Frame: 2 Hours
Population: Response-Evaluable Population 3 with MS, 0 participants in Part A had MS
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Part A | Part B
Number analyzed (Participants) | 0 | 4
percentage
  Brain-Grey Matter |  | 88.339 (10.476)
  Brain-Lesion |  | 73.396 (6.751)
  Brain-White Matter |  | 85.514 (8.202)
  Cerebellum-Grey Matter |  | 88.486 (9.884)
  Cerebellum-White Matter |  | 85.167 (11.593)
  Cerebral Cortex-Grey Matter |  | 88.114 (9.931)
  Cerebral Cortex-White Matter |  | 87.262 (9.439)
  Cerebral Subcortex-Grey Matter |  | 83.233 (9.408)
  Cerebral White Matter-White Matter |  | 79.804 (8.192)

11. Primary Outcome: Percentage of Free Brain BTK Relative to Baseline
Description: Percentage of free brain Burtons Tyrosine Kinase (BTK) relative to baseline
Time Frame: Data Not Collected
Population: Study Terminated, data collection for endpoint did not occur.
Arm/Group | Part A | Part B
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Mean Standardized Uptake Value (SUV) in the Brain
Description: Standardized uptake value (SUV) is Semi-quantitative measurement of tracer uptake in body tissue defined as ratio of radioactivity per unit volume of a region of interest to the radioactivity per unit volume of the whole body.
Time Frame: On visits 1 (Day 1) and vist 2 (2hrs to 6 days after visit 1 tracer administration)
Population: Response-Evaluable 2 Population
Measure: Mean (Standard Deviation); unit: g/mL
Arm/Group | Part A | Part B
Number analyzed (Participants) | 5 | 4
g/mL
  Brain-Grey Matter at visit 1: number analyzed (Participants) | 0 | 3
  Brain-Grey Matter at visit 1 |  | 0.773 (0.101)
  Brain-Grey Matter at visit 2 | 0.606 (0.121) | 0.713 (0.122)
  Brain-Lesion at visit 1: number analyzed (Participants) | 0 | 3
  Brain-Lesion at visit 1 |  | 0.677 (0.103)
  Brain-Lesion at visit 2: number analyzed (Participants) | 0 | 4
  Brain-Lesion at visit 2 |  | 0.623 (0.132)
  Brain-White Matter at visit 1: number analyzed (Participants) | 0 | 3
  Brain-White Matter at visit 1 |  | 0.767 (0.098)
  Brain-White Matter at visit 2 | 0.590 (0.108) | 0.705 (0.122)
  Cerebellum-Grey Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebellum-Grey Matter at visit 1 |  | 0.817 (0.099)
  Cerebellum-Grey Matter at visit 2 | 0.656 (0.135) | 0.755 (0.126)
  Cerebellum-White Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebellum-White Matter at visit 1 |  | 0.857 (0.099)
  Cerebellum-White Matter at visit 2 | 0.672 (0.134) | 0.780 (0.136)
  Cerebral Cortex-Grey Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebral Cortex-Grey Matter at visit 1 |  | 0.763 (0.101)
  Cerebral Cortex-Grey Matter at visit 2 | 0.596 (0.121) | 0.705 (0.122)
  Cerebral Cortex-White Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebral Cortex-White Matter at visit 1 |  | 0.783 (0.101)
  Cerebral Cortex-White Matter at visit 2 | 0.606 (0.118) | 0.725 (0.122)
  Cerebral Subcortex-Grey Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebral Subcortex-Grey Matter at visit 1 |  | 0.797 (0.155)
  Cerebral Subcortex-Grey Matter at visit 2 | 0.674 (0.122) | 0.745 (0.159)
  Cerebral White Matter-White Matter at visit 1: number analyzed (Participants) | 0 | 3
  Cerebral White Matter-White Matter at visit 1 |  | 0.723 (0.084)
  Cerebral White Matter-White Matte at visit 2 | 0.550 (0.096) | 0.658 (0.118)

13. Primary Outcome: Mean Volume of Distribution (VT) in the Brain
Description: Volume of Distribution (VT) is the ratio of the radioligand concentration in a region of interest to the radioligand concentration in plasma at equilibrium.
Time Frame: On visits 1 (Day 1) and vist 2 (2hrs to 6 days after visit 1 tracer administration)
Population: Response-Evaluable 2 Population
Measure: Mean (Standard Deviation); unit: mL/cm³
Arm/Group | Part A | Part B
Number analyzed (Participants) | 5 | 4
mL/cm³
  Brain-Grey Matter at visit 1: number analyzed (Participants) | 0 | 4
  Brain-Grey Matter at visit 1 |  | 2.378 (0.213)
  Brain-Grey Matter at visit 2: number analyzed (Participants) | 4 | 4
  Brain-Grey Matter at visit 2 | 2.498 (0.343) | 2.505 (0.604)
  Brain-Lesion at visit 1: number analyzed (Participants) | 0 | 4
  Brain-Lesion at visit 1 |  | 2.805 (0.680)
  Brain-Lesion at visit 2: number analyzed (Participants) | 0 | 4
  Brain-Lesion at visit 2 |  | 3.095 (1.407)
  Brain-White Matter at visit 1: number analyzed (Participants) | 0 | 4
  Brain-White Matter at visit 1 |  | 2.608 (0.374)
  Brain-White Matter at visit 2: number analyzed (Participants) | 4 | 4
  Brain-White Matter at visit 2 | 2.645 (0.417) | 2.660 (0.677)
  Cerebellum-Grey Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebellum-Grey Matter at visit 1 |  | 2.535 (0.219)
  Cerebellum-Grey Matter at visit 2: number analyzed (Participants) | 4 | 4
  Cerebellum-Grey Matter at visit 2 | 2.715 (0.356) | 2.638 (0.639)
  Cerebellum-White Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebellum-White Matter at visit 1 |  | 2.883 (0.427)
  Cerebellum-White Matter at visit 2: number analyzed (Participants) | 4 | 4
  Cerebellum-White Matter at visit 2 | 2.953 (0.350) | 2.903 (0.822)
  Cerebral Cortex-Grey Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebral Cortex-Grey Matter at visit 1 |  | 2.340 (0.198)
  Cerebral Cortex-Grey Matter at visit 2: number analyzed (Participants) | 4 | 4
  Cerebral Cortex-Grey Matter at visit 2 | 2.453 (0.338) | 2.470 (0.578)
  Cerebral Cortex-White Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebral Cortex-White Matter at visit 1 |  | 2.540 (0.294)
  Cerebral Cortex-White Matter at visit 2: number analyzed (Participants) | 4 | 4
  Cerebral Cortex-White Matter at visit 2 | 2.645 (0.390) | 2.680 (0.660)
  Cerebral Subcortex-Grey Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebral Subcortex-Grey Matter at visit 1 |  | 2.445 (0.315)
  Cerebral Subcortex-Grey Matter at visit 2: number analyzed (Participants) | 4 | 4
  Cerebral Subcortex-Grey Matter at visit 2 | 2.645 (0.404) | 2.710 (0.815)
  Cerebral White Matter-White Matter at visit 1: number analyzed (Participants) | 0 | 4
  Cerebral White Matter-White Matter at visit 1 |  | 2.790 (0.613)
  Cerebral White Matter-White Matte at visit 2: number analyzed (Participants) | 4 | 4
  Cerebral White Matter-White Matte at visit 2 | 2.675 (0.496) | 2.665 (0.712)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: Approximately up to 11 days All-Cause mortality (From randomization to end of study): Approximately up to 11 days
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Part B: BMS-986196 Approximately 370MBq, equivalent to up to 20 μg
Arm/Group | Part A | Part B
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 2/6 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (N=6) | Part B (N=4)
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Clinically significant abnormalities on ECG, VS, laboratory parameters and PE had to be reported as AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT05064436/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT05064436/SAP_001.pdf